CLINICAL TRIAL: NCT00364962
Title: Treatment Result of KTP Laser Nasopharyngectomy in Recurrent NPC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9561703040
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2006-08-16 (Estimated); Status verified 2006-08

CONDITIONS: Recurrent; Nasopharyngeal Carcinoma
Keywords: NPC; Nasopharyngectomy; KTP laser; recurrence
MeSH Terms: conditions — Recurrence; Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Investigate the treatment result of KTP laser nasopharyngectomy in recurrent NPC patients

DETAILED DESCRIPTION:
Nasopharyngeal carcinomas (NPCs) are highly radiosensitive tumors, and the primary treatment of NPCs is radiotherapy.1 Because most patients who have NPC are at advanced stages when initially seen, local failures in terms of persistence or recurrence are not infrequent after primary radiotherapy.2,3 Local regional relapse without the presence of distant failure can still be salvaged and should be aggressively treated. Tumors relapsing in the nasopharynx can be salvaged using either re-irradiation or surgical techniques.1 Although re-irradiation to the recurrent tumor can extent the 5-year actuarial survival rate, it is associated with high morbidity. 4-6 Traditional nasopharyngectomy has been associated with local control rates on the order of 40%~50%, but it has also been associated with complications such as palatal defects, trismus, facial scarring, osteomyelitis, etc.7-10 That is the reason why surgeons continue searching for new methods for performing nasopharyngectomies with lower morbidities.

Nasopharyngectomies are difficult to perform because of the inaccessibility of the nasopharynx. More difficulties are encountered in performing a nasopharyngectomy through the nose due to the restricted surgical field. With advances in techniques of endoscopy and application of the potassium-titanyl-phosphate (KTP) laser in surgery, pathologic lesions located either at the choanal margin or in the nasopharynx can easily be managed with instruments inserted via the nasal cavities. The surgical technique had been accepted by the authority journal. This time, we will review the therapeutic result of KTP-laser nasopharyngectomy in patients with recurrent NPC.

ELIGIBILITY:
Inclusion Criteria:

* recurrent NPC patients

Exclusion Criteria:

* patients with distant metastasis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-04; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ting Tan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan